CLINICAL TRIAL: NCT02052063
Title: Does the Stapled Transanal Rectal Resection (STARR Procedure) Has an Effect on Anal Compliance ?
Acronym: Compli-STARR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013/132/HP
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Rectocele; Intussusception; Surgery; Sphincter Ani Incontinence
Keywords: rectocele; intussusception; surgery
MeSH Terms: conditions — Rectocele; Intussusception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental): Patient who undergone stapled transanal rectal resection for rectocele. Anal compliance will be evaluated before and starting the surgery using endoflip system
  Interventions: Device: stapled transanal rectal resection; Device: Anal compliance measure with Endoflip system

INTERVENTIONS:
Device: stapled transanal rectal resection — transanal rectal resection using staple will be done for rectocele
  Other Names: transanal rectal resection using staple
Device: Anal compliance measure with Endoflip system — Anal compliance will be measured using Endoflip system

SUMMARY:
The stapled transanal rectal resection (STARR) has recently been recommended for patients with obstructed defecation syndrome (ODS) caused by rectocele and rectal wall intussusception.

The aim of STARR is to correct the mechanical outlet obstruction using a stapler device for endorectal resection of the distal rectum.

This technique significantly improves constipation. However, there are several reports of new-onset faecal incontinence after STARR and urgency has been identified as the major side-effect of this procedure.

Although this technique has become an important surgical option in the treatment of obstructive defaecation syndrome, its impact on continence can be problematic and objective data about parameters that predict its result are not yet available One study evaluated the anal function after surgery in 30 patients. In this study, urgency or incontinence was complained by 26% of patients. No sonographically demonstrable sphincter fragmentations were noticed in the endoanal exam performed at the follow-up.

No significant difference was observed in anorectal manometry. Even if data are not statistically significant, resting and squeezing pressures are lower in those patients not satisfied.

Currently, anal canal pressure measurements using ano-rectal manometry are the most common means of assessment of sphincter function. Some studies have been looking at the concept of distending sphincter regions as a better measure of its performance.

The functional lumen imaging probe (FLIP) is a novel technique which has the ability to provide real-time images of the function of human gastrointestinal sphincter during distension. This distensibility technique provides an important new way of studying the anal canal and hence may have a role in testing sphincter competence in patients with disorders after STARR procedure.

Twenty-eight patients will be enrolled in this study over a period of 36 months.

Preoperative assessment will include

* clinical examination
* the Wexner Incontinence Score and the Faecal Incontinence Quality-of-Life Index (FIQL) to rate anal incontinence
* video defecography, anorectal manometry, anal ultrasound (AUS) and measure of anal sphincter distensibility using endoFLIP Follow-up evaluation will scheduled for 3 months after surgery, and will include symptom evaluation (using the same standard questionnaires for incontinence), clinical examination and investigation using anal ultrasound and endoFLIP.

If we demonstrate that this surgical technique can cause anal lesions with decreased sphincter competence, this may lead to a modification of the surgical technique especially in patients at risk of developing postoperative anal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Patient is not under any type of guardianship
* Patient has a rectocele > 3 cm during defecography
* Patient has persistent defecatory troubles despite medical treatment (laxatives for at least 1 month)
* Patient received information and signed the consent form
* Patients having social security coverage

Exclusion Criteria:

* Patient has an asymptomatic rectocele
* Patient with an enterocele at rest upon defecography, with opacification of the small bowel
* Faecal incontinence
* Anal sphincter insufficiency detected by rectal manometry
* Patient with non-rehabilitated anorectal asynchrony
* Patient has previously had rectal surgery or pelvic radiotherapy
* Patient has a anal or rectal lesion, intestinal inflammatory disease
* Anal or rectal tumor
* Immunocompromised subjects
* Positive pregnancy test, by urine
* Psychological condition which would impair participation in the study
* Coagulation disorders
* Patients using anticoagulants
* Participation in any other device or drug study within 30 days prior to enrollment.
* Patient cannot read French
* Patient is under any type of guardianship

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of anal sphincter distensibility | Month 3
  Comparison of anal sphincter distensibility before and 3 months after surgery with cross-sectional area and intra-balloon pressure.
  The device used is Endoflip system

SECONDARY OUTCOMES:
Comparison of Faecal Incontinence Quality-of-Life Index (FIQL) before and 3 months after surgery | Month 3
  Comparison of Faecal Incontinence Quality-of-Life Index (FIQL) before and 3 months after surgery
Comparison of radiological data (Anal ultrasound) | Month 3
  Comparison of radiological data (Anal ultrasound) before and 3 months after surgery Endo-rectal Brüel and Kjaer echographic probe will be used to compare radiological data (conventional endo-rectal echography)
Comparison of Cleveland Clinic Incontinence score (CCIS) before and 3 months after surgery | Month 3
  Comparison between Cleveland Clinic Incontinence score (CCIS)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BRIDOUX, MD, Principal Investigator — UH Rouen
Locations (1):
- UH Rouen, Rouen, France